CLINICAL TRIAL: NCT02041572
Title: Attentional Bias Retraining in Veterans
Acronym: ABR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pacific Islands Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-05/MM/PROMISE 0001
Record Dates: First submitted 2014-01-15; First posted 2014-01-22 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2014-01

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Masking Description: The transition point from the assessment only version of the attention bias program to the retraining/ bias correction version was randomized at the participant level and occurred between weeks 4 and 7 of the 10-week study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Attentional Bias Retraining (Other): Each participant receives 12 sessions. The first three sessions are baseline (assessment only) sessions. The last four sessions must be treatment sessions. The attentional bias intervention starts randomly on sessions 4 - 8, and continues until the end of the 12 sessions.
  Interventions: Behavioral: Attentional bias retraining

INTERVENTIONS:
Behavioral: Attentional bias retraining — Participants complete a computer-based intervention, which is designed to correct cognitive biases associated with PTSD by training to attend to neutral information rather than the trauma-related cue words.

SUMMARY:
The study has two goals. First to develop a computer-based intervention meant to alter cognitive biases that contribute to ongoing PTSD symptoms. Second, we sought to pilot test the intervention in a small sample of veterans for feasibility and acceptability.

DETAILED DESCRIPTION:
Aim 1: Develop Attentional Bias Retraining protocol (Phase 1)

* 1.1 Computerized assessment & retraining programs
* 1.2 Procedures and measures

Aim 2: Implement in pilot sample (Phase 2)

* 2.1: Assess feasibility and tolerability
* 2.2: Collect pilot data to plan future studies
* 2.3: Efficacy estimates based on changes in response time to dot probe task

ELIGIBILITY:
Inclusion Criteria:

* Participated in ground combat operations in Vietnam
* Scored 40 - 80 on PTSD Checklist - Military version
* Availability and willingness to attend 2x weekly computer sessions for 6 weeks

Exclusion Criteria:

* Active substance dependence
* Significant cognitive impairment
* Current and active suicidal or homicidal ideation

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Post-traumatic Checklist - Military version (PCL-M) | Change from Baseline and Post-treatment (1 month after last training session)
  PCL-M assess the 17-cardinal symptoms of PTSD.

SECONDARY OUTCOMES:
Attentional bias scores | Change from Baseline and Post-treatment (1 month after last training session)
  Attentional bias scores represent participants cognitive bias to orient towards trauma-relevant information more quickly than neutral information.

OTHER OUTCOMES:
Daily of PTSD symptoms, specifically hyperarousal and intrusive symptoms (nightmares, reenactments, and triggered and untriggered recall) | Change from Baseline and Post-treatment (1 month after last training session)
  Participants filled out daily symptom log nightly

CONTACTS AND LOCATIONS:
Overall Officials: Margaret-Anne Mackintosh, PhD, Principal Investigator — National Center for PTSD/PHREI
Locations (1):
- National Center for PTSD, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data